CLINICAL TRIAL: NCT02402569
Title: Implantation Feasibility Study of a Multi-electrodes Set for Deep Brain Stimulation in Parkinson Disease (Smart in Vivo 2)
Brief Title: Multi-electrodes Set for Deep Brain Stimulation in Parkinson Disease
Acronym: SIV2
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SIV2
Record Dates: First submitted 2015-01-30; First posted 2015-03-30 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-electrodes / single electrode (Experimental): Multi stimulation / single stimulation
  Interventions: Device: 32 channels Deep Brain Stimulator
- Single-electrode / Multi electrodes (Experimental): Single stimulation / Multi stimulation
  Interventions: Device: 32 channels Deep Brain Stimulator

INTERVENTIONS:
Device: 32 channels Deep Brain Stimulator

SUMMARY:
This study aims to demonstrate innocuity and feasibility of deep brain stimulation with a multi-electrodes set.

DETAILED DESCRIPTION:
Bilateral stimulation in subthalamic nucleus with the multi-electrodes set will be compared with single electrode.

ELIGIBILITY:
Inclusion Criteria:

* more or equal than 18 years old and less than 70 years
* patient affiliated to social security or similarly regime
* informed consent form signed
* parkinson disease (UPDRS III20 score up than 30/108 except for severe tremors)
* motor and non motor dysfunctions
* pre-operative cerebral MRI without lesion
* without chirurgical contraindications
* without psychiatric disease

Exclusion Criteria:

* Pregnant women and lactating mothers
* Ward of court or under guardianship
* Adult unable to express their consent
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent
* Person under legal protection
* Person with carcinological antecedent during precedent 5 years
* Chirurgical or MRI contraindications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Safety, as measured by Number of Participants with Adverse Events | 3 months
  Number of Participants with Adverse Events

SECONDARY OUTCOMES:
Neurologic evaluation | 3 months
  Change in motor and non-motor symptoms assessment with neurologic scales

CONTACTS AND LOCATIONS:
Locations (1):
- CLINATEC, Grenoble, France